CLINICAL TRIAL: NCT00736567
Title: Evaluation of a Diagnostic Enteric Card for Management of Diarrhea in a Clinical Site in Fortaleza, Brazil
Brief Title: Evaluation of a Diagnostic Enteric Card for Management of Diarrhea
Status: Completed | Type: Observational
Sponsor: PATH (Other)
Collaborators: Universidade Federal do Ceara (Other); University of Virginia (Other); Micronics, Inc. (Industry); Washington University Early Recognition Center (Other)
Responsible Party: Sponsor
Other Study IDs: 07-0008; U01AI061187 (NIH)
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2009-09

CONDITIONS: Diarrhea
Keywords: Diarrhea; Diagnostic; Pediatric
MeSH Terms: conditions — Diarrhea; Disease

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Stool samples are retained for future research.
Oversight: Data Monitoring Committee: No

SUMMARY:
PATH is a member of a consortium that is developing a Diagnostic Enterics Card (DEC) which will allow clinicians to diagnose a group of diarrheagenic pathogens linked to morbidity and mortality. The pathogens detected on DEC include Salmonella, Campylobacter jejuni, Shigella species, and Escherichia coli O157:H7. This study will evaluate the performance of the assays and the platform in clinical conditions with non-expert users. It will provide important data on the performance of DEC for at least one target pathogen, an understanding of the potential impact of different sample types on device performance, and human factors associated with instrument interface in the field.

ELIGIBILITY:
Inclusion Criteria:

* Have 3 or greater liquid stools in the past 24 hours.
* Provide written informed consent from at least one parent in the case of children under 18 years of age.
* Provide written informed consent for those participants above 18 years of age.
* Provide assent in the case of children 10 years of age or greater.

Exclusion Criteria:

* Previously enrolled in the study.
* Parents are unwilling or unable to provide written informed consent.
* Report using antibiotics in the last 30 days.
* Adolescent (<18 years old) parent of a child already enrolled in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting with diahrreal symptom to out-patient care facilities in Fortaleza, Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 436 (Actual)
Dates: Start 2008-05; Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Infantil Albert Sabin, Fortaleza, Ceará, Brazil